CLINICAL TRIAL: NCT03349099
Title: The Impact of Ureteral Access Sheath Design on Ease of Placement and Ureteral Wall Injury During Flexible Ureteroscopy
Brief Title: Impact Ureteral Sheath Design During Ureteroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Manoj Monga, MD, Director of Endourology and Stone Disease, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-632
Record Dates: First submitted 2017-11-13; First posted 2017-11-21 (Actual); Results first posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Renal Stone; Nephrolithiasis; Urolithiasis
MeSH Terms: conditions — Nephrolithiasis; Urolithiasis

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Videos will be analyzed by blinded urologists who will rate the extent of ureteral damage on a standardized scale of 0 to 4 according to the study published by Traxer et al. 2013. After the study, subjects will not be contacted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Cook Flexor (Active Comparator): ureteral access sheath
  Interventions: Device: Cook Flexor
- Boston Scientific Navigator HD (Active Comparator): ureteral access sheath
  Interventions: Device: Boston Scientific Navigator

INTERVENTIONS:
Device: Cook Flexor — ureteral access sheath
  Arms: Cook Flexor
Device: Boston Scientific Navigator — ureteral access sheath
  Arms: Boston Scientific Navigator HD

SUMMARY:
The purpose of this study is to assess whether one of two ureteral access sheaths is safer for patients undergoing ureteroscopy. Both sheaths are FDA approved devices and commercially available. The investigators will compare the ability of sheaths to access the kidney through the ureter and will compare damage done to the ureter after completion of the procedure. Access sheaths are standard of care for this procedure; this study seeks to optimize outcomes for patients.

Patients undergoing ureteroscopy who do not have ureteral stents in place and who have not had an ipsilateral procedure within 90 days will be recruited and consented.

DETAILED DESCRIPTION:
The purpose of this study is to compare two ureteral access sheaths in how the sheaths damage the ureter during flexible ureteroscopy.

Condition Intervention Kidney Stones Nephrolithiasis Urolithiasis Device: Cook Flexor or Boston Scientific Navigator HD

Study Type: Interventional Study Design: Intervention Model: Two group randomized assignment Masking: Single blind Primary Purpose: Treatment

Primary Outcome Measures:

• Successful placement of sheath (yes or no).

Secondary Outcome Measures:

* Subjective rating of damage to ureter. At the completion of the procedure, video of the intraluminal ureter is recorded as the sheath is withdrawn. Videos are analyzed by two blinded staff endourologists to score ureteral injury on a standard 5-point scale (0 to 4); reference Traxer and Thomas.
* Ease of placement of each sheath. Surgeons will be asked to subjectively rate the ease of placement on a standardized scale from 0 to 4, 4 being easiest which will be rated by the surgeon who inserted the sheath immediately after placement.

Arms Assigned Interventions Device: Cook Flexor and Boston Scientific Navigator HD Device: Cook Flexor or Boston Scientific Navigator HD Patients will be assigned to one of two ureteral access sheaths. If the first sheath is failed to be placed, the backup sheath will be attempted.

Standard ureteroscopy will take place. The intervention takes place before the ureteral access sheath is placed. The patient will be randomized to one of the two sheaths. The randomized 12/14Fr sheath will be attempted. If placed successfully, the rest of the operation continues as planned. If the initial sheath is unable to be placed, a second backup sheath (opposite brand) will be used, also in size 12/14Fr. The surgeon will be asked to rate the ease of placement of the sheath on a standardized scale. If these sheaths fail, it is the surgeon's discretion to continue with the smaller sheath, continue without sheath or place stents and attempt the procedure at a later date. The operation is then continued in standard fashion. Once the ureteroscopy is completed, before the scope and access sheath are removed, video recording of the ureter will be conducted as the ureteroscopy and sheath are removed.

Videos will be analyzed by blinded urologists who will rate the extent of ureteral damage on a standardized scale of 0 to 4 according to the study published by Traxer et al. 2013. Intra-operative data includes total time of initial sheath insertion (in seconds), total time sheath is in place (minutes) from placement to removal, and use of laser. Differences in operative time, ease of placement, ability to maintain access, and ease of instrument passage are also evaluated between devices, as well as success rates, and device failure rates and post-operative complications. Means are compared using a t-test and proportions are compared using a chi-squared test. An intention to treat model is used for statistical analysis. When video ratings differ between surgeons, the higher rating of damage will be used. Inter-rater reliability is assessed with Cohen's kappa coefficient.

After the study, subjects will not be contacted. The investigators will collect data from participants' medical records including information of whether participants develop complications or return for a subsequent procedure as well as size and location of kidney stones prior to the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for ureteroscopy
* Current CT scan within 90-days before the operation
* Able to give informed consent
* Ages 18 years and older

Exclusion Criteria:

* Inability to give informed consent
* Age less than 18 years
* Pregnant
* Stones in the ureter
* Having previous ipsilateral ureteral or renal surgery within 90 days
* Having stents placed in ipsilateral ureter within 90 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2014-06-27 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manoj Monga, MD, Principal Investigator — Urologist

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kourambas J, Byrne RR, Preminger GM. Does a ureteral access sheath facilitate ureteroscopy? J Urol. 2001 Mar;165(3):789-93. PMID 11176469
- [Background] Rehman J, Monga M, Landman J, Lee DI, Felfela T, Conradie MC, Srinivas R, Sundaram CP, Clayman RV. Characterization of intrapelvic pressure during ureteropyeloscopy with ureteral access sheaths. Urology. 2003 Apr;61(4):713-8. doi: 10.1016/s0090-4295(02)02440-8. PMID 12670551
- [Background] Pietrow PK, Auge BK, Delvecchio FC, Silverstein AD, Weizer AZ, Albala DM, Preminger GM. Techniques to maximize flexible ureteroscope longevity. Urology. 2002 Nov;60(5):784-8. doi: 10.1016/s0090-4295(02)01948-9. PMID 12429296
- [Background] Auge BK, Pietrow PK, Lallas CD, Raj GV, Santa-Cruz RW, Preminger GM. Ureteral access sheath provides protection against elevated renal pressures during routine flexible ureteroscopic stone manipulation. J Endourol. 2004 Feb;18(1):33-6. doi: 10.1089/089277904322836631. PMID 15006050
- [Background] Lallas CD, Auge BK, Raj GV, Santa-Cruz R, Madden JF, Preminger GM. Laser Doppler flowmetric determination of ureteral blood flow after ureteral access sheath placement. J Endourol. 2002 Oct;16(8):583-90. doi: 10.1089/089277902320913288. PMID 12470467
- [Background] Traxer O, Thomas A. Prospective evaluation and classification of ureteral wall injuries resulting from insertion of a ureteral access sheath during retrograde intrarenal surgery. J Urol. 2013 Feb;189(2):580-4. doi: 10.1016/j.juro.2012.08.197. Epub 2012 Oct 8. PMID 22982421
- [Background] Schoenthaler M, Wilhelm K, Kuehhas FE, Farin E, Bach C, Buchholz N, Miernik A. Postureteroscopic lesion scale: a new management modified organ injury scale--evaluation in 435 ureteroscopic patients. J Endourol. 2012 Nov;26(11):1425-30. doi: 10.1089/end.2012.0227. Epub 2012 Aug 27. PMID 22698147
- [Background] Delvecchio FC, Auge BK, Brizuela RM, Weizer AZ, Silverstein AD, Lallas CD, Pietrow PK, Albala DM, Preminger GM. Assessment of stricture formation with the ureteral access sheath. Urology. 2003 Mar;61(3):518-22; discussion 522. doi: 10.1016/s0090-4295(02)02433-0. PMID 12639636
- [Background] Ayyathurai R, Kanagarajah P, Shields J, Young E, Alvarez A, Bird VG. Single-center clinical comparison of two reinforced ureteral access sheaths for retrograde ureteroscopic treatment of urinary lithiasis. Int Urol Nephrol. 2012 Apr;44(2):409-14. doi: 10.1007/s11255-011-0017-8. Epub 2011 Jun 25. PMID 21706214
- [Background] De S, Sarkissian C, Torricelli FC, Brown R, Monga M. New ureteral access sheaths: a double standard. Urology. 2015 Apr;85(4):757-63. doi: 10.1016/j.urology.2014.07.009. Epub 2015 Feb 4. PMID 25661780
- [Background] Mogilevkin Y, Sofer M, Margel D, Greenstein A, Lifshitz D. Predicting an effective ureteral access sheath insertion: a bicenter prospective study. J Endourol. 2014 Dec;28(12):1414-7. doi: 10.1089/end.2014.0215. PMID 25244070
- [Background] Fuganti PE, Pires S, Branco R, Porto J. Predictive factors for intraoperative complications in semirigid ureteroscopy: analysis of 1235 ballistic ureterolithotripsies. Urology. 2008 Oct;72(4):770-4. doi: 10.1016/j.urology.2008.05.042. Epub 2008 Jul 16. PMID 18632141

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted from urology pre-operative clinic from July 1 2014 to May 31 2016
Pre-assignment Details: No patients were excluded prior to assignment.
Period: Overall Study
Arm/Group | Cook Flexor | Boston Scientific Navigator HD
Started | 48 | 47
Completed | 44 | 43
Not Completed | 4 | 4
Not completed — Physician Decision | 3 | 4
Not completed — Stone migrated from the kidney | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cook Flexor | Boston Scientific Navigator HD | Total
Number analyzed (Participants) | 48 | 47 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (9) | 50.4 (11) | 52.1 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 24 | 52
  Male | 20 | 23 | 43
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 48 | 47 | 95

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Sheath Placement
Description: The surgeon documents whether there was Successful placement of sheath (yes or no)
Time Frame: One time point - at the beginning of the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Cook Flexor | Boston Scientific Navigator HD
Number analyzed (Participants) | 44 | 43
Participants | 37 | 39

2. Secondary Outcome: Number of Participants With Injury to the Ureter
Description: Subjective rating of damage to ureter. At the completion of the procedure, video of the intraluminal ureter is recorded as the sheath is withdrawn. Videos are analyzed by two blinded staff endourologists who score ureteral injury on a standard 5-point scale (0 to 4); reference Traxer and Thomas.
Time Frame: One time point - at the completion of the procedure
Population: Patients undergoing procedures with each device.
Measure: Count of Participants; unit: Participants
Arm/Group | Cook Flexor | Boston Scientific Navigator HD
Number analyzed (Participants) | 44 | 43
Participants | 36 | 27

3. Secondary Outcome: Ease of Sheath Placement
Description: Surgeons will be asked to subjectively rate the ease of placement on a standardized scale from 0 to 4, 4 being easiest which will be rated by the surgeon who inserted the sheath immediately after placement.
Time Frame: One time point - at the completion of the procedure
Population: patients undergoing ureteroscopy with each device.
Measure: Number; unit: units on a scale
Arm/Group | Cook Flexor | Boston Scientific Navigator HD
Number analyzed (Participants) | 44 | 43
units on a scale | 2.9 | 3.4

ADVERSE EVENTS:
Time Frame: Data was collected intraoperatively (average time one hour)
Arm/Group | Cook Flexor | Boston Scientific Navigator HD
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/43
Other Adverse Events (participants affected / at risk) | 0/44 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-05-31): https://cdn.clinicaltrials.gov/large-docs/99/NCT03349099/Prot_SAP_000.pdf
  • Informed Consent Form (2014-05-31): https://cdn.clinicaltrials.gov/large-docs/99/NCT03349099/ICF_001.pdf